CLINICAL TRIAL: NCT01260168
Title: Multi-marker Stool Test for Detection of Colorectal Neoplasia: Marker Panel Selection and Technical Development Studies
Status: Completed | Type: Observational
Sponsor: Exact Sciences Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: Exact Sciences 2010-A
Record Dates: First submitted 2010-12-06; First posted 2010-12-15 (Estimated); Last update posted 2015-05-13 (Estimated); Status verified 2015-05

CONDITIONS: Colorectal Neoplasms; Digestive System Diseases; Colonic Diseases; Colorectal Cancer
Keywords: Cancer; Colorectal Cancer; Neoplasm; Colorectal Neoplasm; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Digestive System Diseases; Gastrointestinal Diseases; Colonic Diseases; Intestinal Diseases; Rectal Diseases
MeSH Terms: conditions — Colorectal Neoplasms; Digestive System Diseases; Colonic Diseases; Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Gastrointestinal Diseases; Intestinal Diseases; Rectal Diseases

STUDY DESIGN:
Observational Model: Case-Only
Biospecimen Retention: Samples With DNA — Residual specimens and histopathology tissue slides or blocks will be stored for up to 10 years in the Sponsor's on-site bio-repository or similar commercial bio-repository contracted by the Sponsor.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Colorectal cancer patients: Subjects will be men and women, 40-90 years of age, inclusive, each with a colonoscopic biopsy-based diagnosis of colorectal cancer (CRC) and/or an intact pre-malignant colorectal lesion large enough to require surgical excision or complex colonoscopic polypectomy.

SUMMARY:
The objective of this study is to confirm the sensitivity of a stool DNA test for detection of colorectal cancer and pre-cancer.

Another objective is to provide anonymous, clinically characterized specimens for a bio-repository for future colorectal cancer-related test development.

DETAILED DESCRIPTION:
Patients who have been recently diagnosed with colo-rectal cancer or pre-cancer will be asked to submit a stool sample(s)(at least 7 days AFTER colonoscopy) and will have the option of submitting blood and tissue samples for future colo-rectal cancer-related test development.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is male or female, 40-90 years of age, inclusive.
2. Subject has a diagnosis of CRC, at any stage, confirmed with a tissue biopsy and/or ≥1 cm colorectal polyp/adenoma/mass identified on a colonoscopy that is of sufficient size to require surgical excision or complex colonoscopic polypectomy.
3. Subject understands the study procedures and is able to provide informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Subject has active synchronous extra-colonic aerodigestive tract cancers (e.g., lung, esophagus, stomach, or pancreatic cancer).
2. Subject has a history of any inflammatory bowel disease.
3. Subject has familial adenomatous polyposis, hereditary non-polyposis colorectal cancer (Lynch) syndrome, or other hereditary cancer syndromes.
4. Individual has a condition the Investigator believes would interfere with his or her ability to provide informed consent, comply with the study protocol, which might confound the interpretation of the study results or put the person at undue risk.

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who have had colorectal cancer or pre-malignancy confirmed by colonoscopic biopsy-based diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 435 (Actual)
Dates: Start 2010-10; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
The primary endpoints are point estimates of the sensitivity of the diagnostic tests for detection of colorectal neoplasms. | 12 Months
  The diagnostic test under development is a multi-marker stool test for detecting CRC and pre-cancer in a general screening application. The primary objective of this study is to confirm the sensitivity of the optimal DNA marker panel.

SECONDARY OUTCOMES:
To collect samples from patients diagnosed with colorectal cancers. | 12 Months
  Residual samples from patients diagnosed with colorectal cancer will be archived for further research intended to help in the diagnosis of cancers. Specimens will be stored up to 10 years in the Sponsor's on-site bio-repository or similar commercial bio-repository contracted by the sponsor.

CONTACTS AND LOCATIONS:
Overall Officials: Graham Lidgard, PhD, Study Chair — Chief Scientific Officer
Locations (21):
- United States (20):
  - Achieve Clinical Research, LLC, Birmingham, Alabama
  - Clinical Research Associates, Huntsville, Alabama
  - Atlanta Gastroenterology, Atlanta, Georgia
  - Jesse Brown VA, Chicago, Illinois
  - Rush University Gastroenterologists, Chicago, Illinois
  - Stroger Cook County, Chicago, Illinois
  - University of Illinois at Chicago, Chicago, Illinois
  - Rockford Gastroenterology Associates, Ltd, Rockford, Illinois
  - Gastroenterology Associates, Baton Rouge, Louisiana
  - Chevy Chase Clinical Research, Chevy Chase, Maryland
  - Commonwealth Clinical Studies, Brockton, Massachusetts
  - Long Island Gastrointestinal Group, Great Neck, New York
  - Mount Sinai School of Medicine, New York, New York
  - Asheville Gastroenterology, Asheville, North Carolina
  - Southern Gastroenterology Associates, New Bern, North Carolina
  - Northwest Gastroenterology Clinic, LLC, Portland, Oregon
  - Gastro One, Germantown, Tennessee
  - Digestive Health Specialists, Tyler, Texas
  - University of Utah, Salt Lake City, Utah
  - Digestive and Liver Disease Specialists, Norfolk, Virginia
- University of Calgary, Calgary, Alberta, Canada

REFERENCES:
- [Result] Lidgard GP, Domanico MJ, Bruinsma JJ, Light J, Gagrat ZD, Oldham-Haltom RL, Fourrier KD, Allawi H, Yab TC, Taylor WR, Simonson JA, Devens M, Heigh RI, Ahlquist DA, Berger BM. Clinical performance of an automated stool DNA assay for detection of colorectal neoplasia. Clin Gastroenterol Hepatol. 2013 Oct;11(10):1313-8. doi: 10.1016/j.cgh.2013.04.023. Epub 2013 Apr 29. PMID 23639600